CLINICAL TRIAL: NCT01264302
Title: A Randomized, Single-dose, Two-treatment, Two-way, Crossover Bioequivalence Study of Finasteride 5 mg Tablets (Dr. Reddy's Laboratories Limited) With the Reference Formulation PROSCAR® 5 mg Tablet (Merck & Co., Inc.) Under Fed Conditions in Healthy Adult Male Subjects.
Brief Title: Bioequivalence Study of Two Finasteride 5 mg Tablet Formulations Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sr. Director- Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10640610
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2006-12

CONDITIONS: Healthy
Keywords: Bioequivalence; Finasteride; crossover
MeSH Terms: interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Finasteride tablets 5 mg (Experimental): Finasteride tablets 5 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Finasteride
- Proscar 5 mg Tablets (Active Comparator): Proscar 5 mg Tablets of Merck & Co. Inc
  Interventions: Drug: Finasteride

INTERVENTIONS:
Drug: Finasteride — Finasteride Tablets 5 mg
  Other Names: Proscar

SUMMARY:
The objective of this study was to evaluate the relative bioavailability of the test formulation of finasteride 5 mg tablets (Dr. Reddy's Laboratories Limited) with the reference formulation PROSCAR® 5 mg Tablet (Merck & Co., Inc.)under fed conditions in healthy adult male subjects.

DETAILED DESCRIPTION:
This randomized, single-dose, two-treatment, two-way, crossover study was conducted to compare the relative bioavailability of two formulations of 5 mg finasteride tablets under fed conditions. The study was conducted with 26 (24 completed) healthy adults. The subjects received the test product in one study period and the reference product in the other period; the order of administration was according to the dosing randomization schedule. There was a 7-day interval between treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Males, 18-65 years of age (inclusive).
2. A body mass index (BMI) of 18-30 kg/m2 inclusive as calculated according to Novum Standard Operating Procedures.
3. Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
4. Signed and dated informed consent form, which meets all criteria of current FDA regulations.

Exclusion Criteria:

1. Female.
2. History of allergy or sensitivity to finasteride, or similar drugs, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
3. Significant history or current evidence of chronic infectious disease, system disorder or organ dysfunction.
4. Presence of gastrointestinal disease or history of malabsorption within the last year.
5. History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
6. Presence of a medical condition requiring regular treatment with prescription drugs.
7. Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to initial dosing.
8. Receipt of any drug as part of a research study within 30 days prior to dosing.
9. Drug or alcohol addiction requiring treatment in the past 12 months.
10. Donation or significant loss of whole blood (480 ml or more) within 30 days or plasma within 14 days prior to dosing.
11. Positive test results for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
12. Positive test results for drugs of abuse at screening.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-11; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Darin B. Brimhall, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Las Vegas, Nevada, United States